CLINICAL TRIAL: NCT05755750
Title: Clinical and Ultrasonographic Evaluation of Intratendinous Genipin Injection in Horses With Superficial Digital Flexor Tendon Injuries
Brief Title: Intratendinous Genipin Injection in Horses With Tendon Injuries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Corsin Heim, Dr. med. vet., University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genipin
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Superficial Digital Flexor Tendonitis
MeSH Terms: interventions — genipin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratendinous genipin injection (Experimental): Genipin was administrated intratendinously under sonographic guidance. For lesions up to 3 cm in length, two separate 0.2 ml injections of genipin solution were administered into the region of transition from degenerated to normal tendon tissue. One injection was given at the proximal end of the lesion and the other at the distal end.
  For lesions longer than 3 cm, an additional 0.2 ml injection was used for every additional 3 cm of lesion length. In the illustrated example, the 6 cm lesion required a total of three injections, and therefore one additional injection was given in the middle of the lesion between the distal and proximal injections.
  Genipin treatment solution contained 100 mM genipin and 20% of the solvent dimethyl sulfoxidee in phosphate buffered saline. Instead of one administration of a relatively large volume, several individual administrations of 0.2 ml were performed depending on lesion size .
  Interventions: Drug: Genipin

INTERVENTIONS:
Drug: Genipin — Intratendinous genipin injection
  Other Names: Methyl (1R,4aS,7aS)-1-hydroxy-7-(hydroxymethyl)-1,4a,5,7a-tetrahydrocyclopenta[c]pyran-4-carboxylate

SUMMARY:
Our study is the first to use genipin, a naturally occurring collagen cross-linking agent, as a therapeutic agent to treat superficial digital flexor tendon (SDFT) injuries in horses. The promising approach of intratendinous genipin injection and tendon mechanical enhancement could be a viable alternative to current therapies for SDFT injuries.

DETAILED DESCRIPTION:
Tendon injuries are a career limiting or ending condition in horses. Genipin (GP), an exogenous collagen crosslinker, provides ex-vivo tendon mechanical augmentation and excellent biosafety. The main objective of this study is to investigate treatment success of GP-induced collagen crosslinking in a clinical application in horses with superficial digital flexor tendon (SDFT) injuries. Horses with an AAEP (American Association of American Practitioners) lameness score > 0 and sonographically confirmed tendinopathy are treated with intratendinous GP injection (IGI) and controlled exercise. Minimal follow-up was set at 12 months. Outcome factors are lameness (AAEP lameness score), soundness, assessment of return to previous use, and re-injury. Additionally, adverse effects are recorded.

ELIGIBILITY:
Inclusion Criteria:

* clinical and sonographic evidence of a tendon injury

Exclusion Criteria:

* in the final analysis, only superficial digital flexor tendon injuries were included
* if follow-up was less than 12 m due to euthanasia, death or other reasons, horses were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Recovery from tendon injury | 12 months
  The amount of horses that regain AAEP lameness grade 0 (sound; free of lameness) after superficial digital flexor tendon injury

CONTACTS AND LOCATIONS:
Overall Officials: Fürst Anton, Prof Dr., Study Director — Professor, Head of Department
Locations (1):
- Equine surgery, Vetsuisse-Faculty, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No